CLINICAL TRIAL: NCT00794274
Title: The Efficacy and Safety of CC-10004 in Chronic Cutaneous Sarcoidosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Celgene Corporation (Industry); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Robert P Baughman, Professor of Medicine, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP0005
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Sarcoidosis; Cutaneous Sarcoidosis
Keywords: Sarcodiosis; tumor necrosis factor
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label drug (Experimental): Drug: CC-100004
  After the screening period, subjects will receive CC-10004 20mg by mouth BID for 84 days. The 84-day duration of treatment is expected to provide adequate time to assess the short-term efficacy and safety of CC-10004 in a population of subjects with chronic cutaneous sarcoidosis
  Interventions: Drug: CC-100004

INTERVENTIONS:
Drug: CC-100004 — After the screening period, subjects will receive CC-10004 20mg by mouth BID for 84 days. The 84-day duration of treatment is expected to provide adequate time to assess the short-term efficacy and safety of CC-10004 in a population of subjects with chronic cutaneous sarcoidosis.
  Other Names: Aprelimast

SUMMARY:
To determine whether CC-10004, a phosphodiesterase inhibitor, is useful in treating chronic cutaneous sarcoidosis.

DETAILED DESCRIPTION:
This will be an open label, phase II trial of CC-10004 for chronic cutaneous sarcoidosis. It will include two centers (University of Cincinnati and Medical University of South Carolina). The study will evaluate patients with chronic disease who are on a stable treatment regimen and have no significant change in their Sarcoidosis Skin Activity and Severity Index score (SASI) at two visits at least one month apart.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form
* Must be male or female and aged ≥ 18 years at time of consent
* Must be able to adhere to the study visit schedule and other protocol requirements
* Patients with sarcoidosis as defined by the ATS/ERS/WASOG statement on sarcoidosis as defined by the clinical presentation consistent with sarcoidosis, biopsy finding granulomas, and no alternative for the cause of the granulomas, such as tuberculosis
* Patients must have chronic cutaneous skin lesions while taking chronic therapy (corticosteroids, methotrexate (max 10mg/week), azathioprine, hydroxychloroquine, cyclophosphamide, minocycline, doxycycline and chloroquine), in which the dose has not been altered in the three months prior to starting the study.
* Must have two visits within the previous 1-6 months (at least one month apart) with stable skin lesions, such as a SASI score was within one point for each of the features of the lesion.
* Must meet the following laboratory criteria:

  * Hemoglobin > 9 g/dL
  * Hematocrit ≥ 27%
  * White blood cell (WBC) count ≥ 3000 (≥ 3.0 X 109/L) and < 20,000 (< 20 X 109/L)
  * Neutrophils ≥ 1500 (≥ 1.5 X 109/L)
  * Platelets ≥ 100,000 (≥ 100 X 109/L)
  * Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L)
  * Total bilirubin < 2.0 mg/dL
  * Aspartate transaminase (AST [serum glutamic oxaloacetic transaminase, SGOT]) and alanine transaminase (ALT [serum glutamate pyruvic transaminase, SGPT]) < 1.5x upper limit of normal (ULN)
* Females of childbearing potential (FCBP)‡ must have a negative urine pregnancy test at screening (Visit 1). In addition, sexually active FCBP must agree to use TWO of the following adequate forms of contraception while on study medication: oral, injectable, or implantable hormonal contraceptives; tubal ligation; intrauterine device; barrier contraceptive or vasectomized partner. A FCBP must agree to have pregnancy tests every 28 days while on study medication.
* Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in sexual activity with FCBP while on study medication and for 84 days after taking the last dose of study medication.

Exclusion Criteria:

* History of any clinically significant cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic, or other major diseases (not including pulmonary sarcoidosis)
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Pregnant or lactating female
* History of active Mycobacterium tuberculosis infection (any subspecies) within 3 years prior to the screening visit. Infections that occurred > 3 years prior to entry must have been effectively treated.
* History of incompletely treated latent Mycobacterium tuberculosis infection (as indicated by a positive Purified Protein Derivative [PPD] skin test or in vitro test [T-SPOT®.TB, QuantiFERON Gold®].
* Clinically significant abnormality on the chest x-ray (CXR) at screening not due to sarcoidosis
* Use of any investigational medication within 28 days.
* Any clinically significant abnormality on 12-lead ECG at screening
* Positive human immunodeficiency virus (HIV), hepatitis B, or hepatitis C laboratory test result indicating active infection at screening
* History of malignancy within previous 5 years (except for treated basal-cell skin carcinoma(s) and/or fewer than 3 treated squamous-cell skin carcinomas)
* Use of infliximab, etanercept, adalimumab, pentoxifylline, or thalidomide in the prior three months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Improvement in skin lesions as assessed by a Sarcoidosis Skin Activity and Severity Index (SASI) . | 6 months

SECONDARY OUTCOMES:
To determine the safety (type, frequency, severity, and relationship of adverse events to study treatment) of CC-10004 in patients with chronic cutaneous sarcoidosis. | 6 months
Improvement of global score of sarcoidosis using a visual analogue scale (VAS) by both the patient and a separate VAS by the physician. | 6 months
Change in the quality of life using the Sarcoidosis Health Questionnaire and Short Form-36 (SF-36). | 6 months
Change in genomic and proteomic expression of cytokines in paired skin biopsies (non-facial lesions). | 6 months
Improvement in pulmonary status, specifically the six-minute walk test, dyspnea score, and forced vital capacity (FVC). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Baughman, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Baughman RP, Judson MA, Ingledue R, Craft NL, Lower EE. Efficacy and safety of apremilast in chronic cutaneous sarcoidosis. Arch Dermatol. 2012 Feb;148(2):262-4. doi: 10.1001/archdermatol.2011.301. Epub 2011 Oct 17. No abstract available. PMID 22004880